CLINICAL TRIAL: NCT03643575
Title: A Phase I, Open- Label, Randomized, Multiple-dose, 3-way Crossover Relative Bioavailability Study to Characterize the Pharmacokinetics of the 3 Marketed Products Containing 200 mg Guaifenesin Under Fasted Conditions in Normal Healthy Subjects.
Brief Title: Study to Characterize the Pharmacokinetics of 3 Marketed Products Containing 200 mg Guaifenesin in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Inc. (Industry)
Responsible Party: Sponsor
Organization: Reckitt Benckiser LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-GGE-05
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Results first posted 2019-02-22 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment A: Vicks Cough Syrup for Chesty Coughs (Experimental): Vicks Cough immediate-release (IR) syrup 15 mL (containing 200 mg guaifenesin) every 4 hours x 3 doses with 240 mL of water after an overnight fast
  Interventions: Drug: Vicks Cough Syrup for Chesty Coughs
- Treatment B: Robitussin Extra Strength Chest Congestion (Experimental): Robitussin Extra Strength Chest Congestion 5 ml (containing 200 mg guaifenesin) every 4 hours x 3 doses with 240 mL of water after an overnight fast
  Interventions: Drug: Robitussin Extra Strength Chest Congestion
- Treatment C: Organ-I- NR tablet (Experimental): Organ-I- NR 200 mg guaifenesin tablet every 4 hours x 3 doses with 240 mL of water after an overnight fast
  Interventions: Drug: Organ-I- NR tablet

INTERVENTIONS:
Drug: Vicks Cough Syrup for Chesty Coughs — Vicks Cough Syrup for Chesty Coughs 15 mL (containing 200 mg guaifenesin) IR syrup with 240 mL of water
  Arms: Treatment A: Vicks Cough Syrup for Chesty Coughs
Drug: Robitussin Extra Strength Chest Congestion — Robitussin Extra Strength Chest Congestion 5 mL (containing 200 mg guaifenesin) IR syrup with 240 mL of water
  Arms: Treatment B: Robitussin Extra Strength Chest Congestion
Drug: Organ-I- NR tablet — Organ-I- NR tablet (containing 200 mg guaifenesin) with 240 mL of water
  Arms: Treatment C: Organ-I- NR tablet

SUMMARY:
Characterize the relative pharmacokinetics (PK) of 3 marketed products containing guaifenesin

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females between the ages of 19 and 55 years, inclusive.
2. Females of childbearing potential must be using one of the following acceptable birth control methods:

   1. Intra-uterine device in place for at least 3 months prior to Day 1 of Period 1 through 30 days beyond study completion;
   2. Barrier method (condom or diaphragm) with spermicide for at least 7 days prior to screening through 30 days beyond study completion;
   3. Stable hormonal contraceptive (e.g., oral, depo injection, transdermal patch, or vaginal ring) for at least 3 months prior to Day 1 of Period 1 through 30 days beyond completion of study;

   Abstinence is not an acceptable form of contraception; however, abstinent female subjects may be admitted to the study if they agree, and have signed a statement to the effect, that upon becoming sexually active, will use a condom with spermicide from screening through 30 days beyond completion of the study.
3. Females of non-childbearing potential should be surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to study or hysterectomy and/or bilateral oophorectomy at least 3 months prior to Day 1 of Period 1) or postmenopausal >2 years prior to Day 1 of Period 1. A follicle stimulating hormone (FSH) concentration >40 miU/mL must be obtained and recorded for any postmenopausal females.
4. Good general health as determined by the Principal Investigator's (PI) review of medical history, physical examination, vital sign measurements, electrocardiogram (ECG), and clinical laboratory measures.
5. Within 15% of ideal body weight (Table of 'Desirable Weights of Adults' Metropolitan Life Insurance Company, 1983).
6. Non-tobacco users, who have not used nicotine or nicotine-containing products for at least 365 days prior to Day 1 of Period 1.
7. Able to read, understand and sign the informed consent after the nature of the study has been explained.
8. Negative urine screen for drugs of abuse and alcohol at screening and each check in.
9. If female, negative finding on serum pregnancy test at screening and each check-in.

Exclusion Criteria:

1. Clinically significant abnormalities detected by medical history, physical examination, vial sign measurements, ECG, or clinical laboratory findings (as determined by the PI/designee) including a hemoglobin value <12 g/dL at screening. If a subject's hemoglobin drops below 11.0 g/dL during the study, the subject may be dropped from the study at the discretion of the PI.
2. Any disease or condition, which could impact absorption, distribution, metabolism, or elimination of the study drugs (as determined by the PI/designee).
3. Alcoholism or medicinal product or drug abuse within the past two years or excessive alcohol consumption (more than 10 units per week) (one unit is defined as 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of spirits (i.e., 'hard' liquor such as gin, whiskey, or vodka, et. al.). The subject is not to experience tolerance, withdrawal, compulsive use, or substance related problems such as medical complications, disruption in social and family relationships, vocational or financial difficulties, or legal problems.
4. Females who are pregnant or nursing.
5. History of sensitivity reaction to guaifenesin.
6. History of or intolerance to lactose.
7. Receipt of an investigational drug within 30 days prior to Day 1 of Period 1.
8. Abnormal diet (for whatever reason) during the 30 days prior to Day 1 of Period 1.
9. Donation of blood or significant loss of blood within 56 days or plasma within 14 days prior to Day 1 of Period 1.
10. Known or suspected use of illicit drugs.
11. The use of any medication (with the exception of hormonal contraceptives for women of childbearing potential) for 14 days or 5 half-lives of the drug (whichever is longer) prior to Day 1 of Period 1, if not approved by Investigator.
12. Test positive for Hepatitis B surface antigen, Hepatitis C antibodies, or HIV at Screening.
13. Subjects who have participated in previous Reckitt Benckiser studies.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2009-07-16 (Actual); Study Completion 2009-07-16 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study.
Pre-assignment Details: A total of 30 subjects entered the study, among them 27 subjects completed the study.
Groups:
- Treatment Sequence 1: Period 1: Treatment A
  Vicks Cough Syrup 15ml containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 2: Treatment B
  Robitussin Extra Strength 5mL syrup containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 3: Treatment C
  Organ-I NR Tablet containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  There was a 7 days washout period between each administration
- Treatment Sequence 2: Period 1: Treatment B
  Robitussin Extra Strength 5ml syrup containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 2: Treatment C
  Organ-I NR Tablet containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 3: Treatment A
  Vicks Cough Syrup 15ml containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  There was a 7 days washout period between each administration
- Treatment Sequence 3: Period 1: Treatment C
  Organ-I NR Tablet containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 2: Treatment A
  Vicks Cough Syrup 15 mL containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 3: Treatment B
  Robitussin Extra Strength 5mL syrup containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  There was a 7 days washout period between each administration
- Treatment Sequence 4: Period 1: Treatment A
  Vicks Cough Syrup 15 mL containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 2: Treatment C
  Organ-I NR Tablet containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 3: Treatment B
  Robitussin Extra Strength 5mL syrup containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  There was a 7 days washout period between each administration
- Treatment Sequence 5: Period 1: Treatment B
  Robitussin Extra Strength 5mL syrup containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 2: Treatment A
  Vicks Cough Syrup 15 mL containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 3: Treatment C
  Organ-I NR Tablet containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  There was a 7 days washout period between each administration
- Treatment Sequence 6: Period 1: Treatment C
  Organ-I NR Tablet containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 2: Treatment B
  Robitussin Extra Strength 5mL syrup containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Period 3: Treatment A
  Vicks Cough Syrup 15 mL containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  There was a 7 days washout period between each administration
Period: Period 1
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout: 7 Days
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 4 | 5 | 5
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrew consent due to illness | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 4 | 5 | 5 | 4 | 5 | 5
Completed | 4 | 5 | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout: 7 Days
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 4 | 5 | 5 | 4 | 5 | 5
Completed | 4 | 4 | 5 | 4 | 5 | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Non compliance check in | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 4 | 4 | 5 | 4 | 5 | 5
Completed | 4 | 4 | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Treatment A:
  Vicks Cough Syrup 15 mL containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Treatment B:
  Robitussin Extra Strength 5mL syrup containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  Treatment C:
  Organ-I NR Tablet containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
  There was a 7 days washout period between each administration
  Participants randomized to receive either Treatment A or Treatment B or Treatment C in 3 Periods (Period 1, 2, 3) of 6 sequence (ABC, BCA, CAB, ACB, BAC, CBA)
Arm/Group | Overall Study
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race [Number; unit: participants]
  Asian | 1
  Black | 1
  Caucasian | 25
  European/Middle Eastern | 1
  Hispanic | 2
Weight [Mean (Standard Deviation); unit: lb] | 157.60 (22.359)
Height [Mean (Standard Deviation); unit: in] | 69.65 (3.246)
Frame Size [Number; unit: participants]
  Small | 4
  Medium | 23
  Large | 3
Elbow Breadth [Mean (Standard Deviation); unit: in] | 2.661 (0.2140)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Guaifenesin
Description: Pharmacokinetic Parameter Cmax is the Maximum observed plasma concentration.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: Pharmacokinetic (PK) analyses were performed on the available data of the subjects that completed at least 1 period.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment A: Vicks Cough Syrup 15 mL containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
- Treatment B: Robitussin Extra Strength 5mL syrup containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
- Treatment C: Organ-I NR Tablet containing 200 mg guaifenesin every 4 hour for 3 doses by mouth after an overnight fast
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
ng/mL | 1730 (723) | 1230 (456) | 1110 (433)

2. Primary Outcome: Maximum Measured Plasma Concentration at Steady State (Cmax,ss) of Guaifenesin Following the Third Dose
Description: Pharmacokinetic Parameter Cmax,ss is the Maximum observed plasma concentration following the third dose.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
ng/mL | 876 (548) | 765 (309) | 796 (317)

3. Primary Outcome: Observed Plasma Concentration at the End of Dosing Interval at Steady State (Cmin,ss) of Guaifenesin Following the Third Dose
Description: Observed plasma concentration at the end of the dosing interval following the third dose (that is, 4 hours following the third dose).
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
ng/mL | 60.3 (33.4) | 55.1 (28.0) | 73.6 (59.9)

4. Primary Outcome: Average Plasma Concentration (Cav) of Guaifenesin Following the Third Dose
Description: Average plasma concentration (Cav) following the third dose, calculated as AUC(8-12) divided by the dosing interval, 4.
  Cav is calculated as AUC(8-12) / dosing interval, 4
Time Frame: 8, 8.5, 8.75, 9, 9.5, 10, 11 and 12 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
ng/mL | 357 (168) | 313 (128) | 300 (128)

5. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Guaifenesin
Description: Pharmacokinetic Parameter Tmax is the time of the maximum observed plasma concentration.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
hr | 2.66 (2.32) | 2.94 (2.00) | 3.91 (2.29)

6. Primary Outcome: Time to Maximum Observed Plasma Concentration at Steady State (Tmax,ss) of Guaifenesin Following the Third Dose
Description: Pharmacokinetic Parameter Tmax, ss is the time of the maximum observed plasma concentration following the third dose.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
hr | 8.70 (0.333) | 8.67 (0.244) | 9.02 (0.374)

7. Primary Outcome: Apparent First-order Terminal Elimination Half-life (T1/2) of Guaifenesin
Description: T1/2 is the apparent first-order terminal elimination half-life, calculated as ln(2)/Kel.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 27 | 28
hr | 0.961 (0.0973) | 1.04 (0.138) | 0.941 (0.130)

8. Primary Outcome: Apparent First-order Terminal Elimination Rate Constant (Kel) of Guaifenesin
Description: Kel is the apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares (LS) regression analysis using the maximum number of points (e.g., 3 or more non-zero plasma concentrations) in the terminal log-linear phase.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 27 | 28
1/hr | 0.729 (0.0780) | 0.677 (0.0898) | 0.750 (0.0987)

9. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Measurable Concentration [AUC(0-t)] of Guaifenesin
Description: AUC(0-t) is the area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration, as calculated by the linear trapezoidal method.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
ng*hr/mL | 5588.99 (2329.08) | 4369.98 (1708.25) | 4223.74 (1798.98)

10. Primary Outcome: Area Under Plasma Concentration Versus Time Curve From Time 0 to Infinity [AUC(0-inf)] of Guaifenesin
Description: AUC(0-inf) is the area under the plasma concentration versus time curve from time 0 to infinity, calculated as AUC(0-t) + Ct/Kel, where Ct was the last measurable concentration and Kel is the apparent first-order terminal elimination rate constant.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 27 | 28
ng*hr/mL | 5596.33 (2330.20) | 4427.06 (1721.91) | 4232.61 (1801.69)

11. Primary Outcome: Area Under Plasma Concentration Versus Time Curve From 0 to 4 Hours [AUC(0-4)] of Guaifenesin
Description: AUC(0-4) is the area under the plasma concentration versus time curve from time 0 to 4 hours post dose (relative to first dose), as calculated by the linear trapezoidal method.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3 and 4 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
ng*hr/mL | 2013.16 (785.006) | 1490.15 (579.667) | 1414.18 (617.126)

12. Primary Outcome: Area Under Plasma Concentration Versus Time Curve From Time 8 to 12 Hours [AUC(8-12)] of Guaifenesin
Description: AUC(8-12) is the area under the plasma concentration versus time curve from time 8 to 12 hours postdose (relative to first dose), as calculated by the linear trapezoidal method.
Time Frame: 8, 8.5, 8.75, 9, 9.5, 10, 11 and 12 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
ng*hr/mL | 1427.70 (672.821) | 1253.09 (511.519) | 1198.55 (511.210)

13. Primary Outcome: Area Under Plasma Concentration Curve Ratio (AUCR) of Guaifenesin
Description: Pharmacokinetic Parameter AUCR is the Ratio of AUC(0-t) to AUC(0-inf). AUCR = AUC(0-t) / AUC(0-inf).
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 27 | 28
Ratio | 0.9986 (0.000592) | 0.9982 (0.001138) | 0.9978 (0.001724)

14. Primary Outcome: Accumulation Index (AI) of Guaifenesin
Description: AI is the accumulation index, calculated as AUC(8-12) / AUC(0-4).
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4 hours and 8, 8.5, 8.75, 9, 9.5, 10, 11, 12 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
Ratio | 0.7056 (0.1299) | 0.8420 (0.1180) | 0.8592 (0.1304)

15. Primary Outcome: Degree of Fluctuation (DF) of Guaifenesin
Description: DF is the Degree of Fluctuation Index, calculated as (Cmax,ss - Cmin,ss) / Cav.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: Percent fluctuation in concentration
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
Percent fluctuation in concentration | 2.220 (0.5508) | 2.312 (0.5221) | 2.463 (0.6758)

16. Primary Outcome: Peak Plasma Concentrations at Steady State (Swing) of Guaifenesin
Description: Pharmacokinetic Parameter Swing is Calculated as (Cmax,ss - Cmin,ss) / Cmin,ss.
Time Frame: 0 (Pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 4.5, 4.75, 5, 5.5, 6, 7, 8, 8.5, 8.75, 9, 9.5, 10, 11, 12, 14 and 16 hours
Population: PK analyses
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 26 | 28 | 28
Percentage | 16.19 (10.03) | 15.62 (8.908) | 0.750 (0.0987)

17. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Intensity was determined by the Investigator. For symptomatic Adverse Events (AEs) the following definitions were applied.
  Mild = AE did not limit usual activities; subject may have experienced slight discomfort.
  Moderate = AE resulted in some limitation of usual activities; subject may have experienced significant discomfort.
  Severe = AE resulted in an inability to carry out usual activities; subject may have experienced intolerable discomfort/pain.
  Relationship to Investigational Medicinal Products (IMP)
  Unlikely = Slight, but remote, chance that AE was caused by IMP. Possible = Reasonable suspicion that the AE was caused by IMP. Probable = Most likely that AE was caused by IMP.
Time Frame: Up to day 2 (Period 3)
Population: PK analyses
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 29 | 28 | 28
participants
  TEAE by severity: Mild | 5 | 1 | 4
  TEAE by severity: Moderate | 2 | 0 | 1
  TEAE by severity: Severe | 0 | 0 | 0
  Relationship to IMP - Unlikely | 5 | 1 | 2
  Relationship to IMP - Possible | 1 | 0 | 2
  Relationship to IMP - Probable | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to day 2 (Period 3)
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 5/29 | 1/28 | 4/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=29) | Treatment B (N=28) | Treatment C (N=28)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No